CLINICAL TRIAL: NCT04419389
Title: Phase 1 and Dose Expansion Study of APR-246 in Combination With Acalabrutinib or Venetoclax-based Therapy in Subjects With R/R NHL Including Chronic Lymphocytic Leukemia (CLL) and Mantle Cell Lymphoma (MCL)
Brief Title: APR-246 in Combination With Acalabrutinib or Venetoclax Based Therapy in Subjects With R/R Non Hodgkin Lymphomas (NHL)
Acronym: R/R
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Aprea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A20-11197
Record Dates: First submitted 2020-06-01; First posted 2020-06-05 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Non Hodgkin Lymphoma; Chronic Lymphocytic Leukemia; Mantle Cell Lymphoma
Keywords: APR-246; eprenetapopt
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell | interventions — eprenetapopt; acalabrutinib; venetoclax; Rituximab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Safety Lead-In Cohort 1 (Experimental): APR-246 4.5 g/d + Acalabrutinib in Subjects with R/R CLL (APR 246 Monotherapy Lead-in; 4.5 g/d x 2)
  Interventions: Drug: APR-246 (eprenetapopt) + Acalabrutinib in CLL
- Safety Lead-In Cohort 2 (Experimental): APR-246 4.5 g/d + Venetoclax + Rituximab in Subjects with R/R CLL (APR 246 Monotherapy Lead-in; 4.5 g/d x 2).
  Interventions: Drug: APR-246 (eprenetapopt) 4.5 g/d + Venetoclax + Rituximab in CLL
- Expansion Cohorts (Experimental): APR-246 4.5 g/d + (Acalabrutinib, OR, (Ven+R)) in Subjects with R/R TP53-mutant CLL, and/or MCL, and/or RT
  Interventions: Drug: APR-246 (eprenetapopt) 4.5 g/d + (Acalabrutinib, OR, (Venetoclax +Rituximab)), in CLL and/or MCL and/or RT
- Safety Lead-In Cohort 3 (Experimental): APR-246 4.5 g/d + Venetoclax + Rituximab in Subjects with RT
  Interventions: Drug: APR-246 (eprenetapopt) 4.5 g/d + Venetoclax + Rituximab in RT

INTERVENTIONS:
Drug: APR-246 (eprenetapopt) + Acalabrutinib in CLL — APR-246 D1, 8 and 15 of each cycle Acalabrutinib will be given at a standard dose and schedule (APR 246 Monotherapy Lead-in; 4.5 g/d x 2)
  Arms: Safety Lead-In Cohort 1
Drug: APR-246 (eprenetapopt) 4.5 g/d + Venetoclax + Rituximab in CLL — APR-246 D1, 8 and 15 of each cycle Venetoclax + Rituximab will be given at a standard dose and schedule (APR 246 Monotherapy Lead-in; 4.5 g/d x 2)
  Arms: Safety Lead-In Cohort 2
Drug: APR-246 (eprenetapopt) 4.5 g/d + (Acalabrutinib, OR, (Venetoclax +Rituximab)), in CLL and/or MCL and/or RT — APR-246 D1, 8 and 15 of each cycle Acalabrutinib will be given at a standard dose and schedule Venetoclax and Rituxiab will be given at a standard dose and schedule
  Arms: Expansion Cohorts
Drug: APR-246 (eprenetapopt) 4.5 g/d + Venetoclax + Rituximab in RT — APR-246 4.5 g/d D1, 8 and 15 of each cycle Venetoclax + Rituximab will be given at a standard dose and schedule
  Arms: Safety Lead-In Cohort 3

SUMMARY:
Study to determine the preliminary safety, tolerability, and pharmacokinetic (PK) profile of APR-246 in combination with either acalabrutinib or venetoclax + rituximab therapy in subjects with NHL, including relapsed and/or refractory (R/R) CLL and R/R MCL.

DETAILED DESCRIPTION:
Phase 1, open-label, dose-finding and cohort expansion study to determine the preliminary safety, tolerability, and pharmacokinetic (PK) profile of APR-246 (eprenetapopt) in combination with either acalabrutinib or venetoclax + rituximab therapy in subjects with NHL, including relapsed and/or refractory (R/R) CLL and R/R MCL.

The study includes a safety lead-in portion followed by an expansion portion in subjects with R/R CLL, Richter Transformation (RT), and R/R MCL.

ELIGIBILITY:
Inclusion Criteria:

1. Is able to understand and is willing and able to comply with the study requirements and to provide written informed consent.
2. Documented histologic diagnosis of R/R CLL, RT, or R/R MCL
3. Safety Lead-In Cohort 1: Patients whose most recent regimen did not include BTK inhibitor therapy.
4. Safety Lead-In Cohort 2: Patients whose most recent regimen did not include Bcl-2 inhibitor therapy.
5. Safety Lead-In Cohort 3: APR-246 + venetoclax + rituximab in patients with RT
6. Prothrombin time (or international normalized ratio) and partial thromboplastin time not to exceed 1.2 × the institution's normal range.
7. Adequate BM function independent of growth factor or transfusion support, per local laboratory reference range at screening as follows:

   1. platelet count ≥ 75 000/mm3;
   2. absolute neutrophil count (ANC) ≥ 1000/mm3 unless cytopenia is clearly due to marrow involvement from CLL or MCL
   3. total hemoglobin ≥ 9 g/dL (without transfusion support within 2 weeks of screening);
8. Adequate organ function as defined by the following laboratory values:

   1. Creatinine clearance ≥ 30 mL/min.
   2. Total serum bilirubin ≤ 1.5 × upper limit of normal (ULN) unless due to Gilbert's syndrome, NHL organ involvement, controlled immune hemolysis or considered an effect of regular blood transfusions.
   3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN, unless due to NHL organ involvement.
9. Age ≥18 years at the time of signing the informed consent form.
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
11. Projected life expectancy of ≥ 12 weeks.
12. Women of childbearing potential and men with female partners of childbearing potential must be willing to use an effective form of contraception.

    Exclusion Criteria:
13. Patient with known allergies to xanthine oxidase inhibitors and/or rasburicase.
14. For patients to receive rituximab on this protocol, prior allergy to rituximab is prohibited.
15. No concomitant anticancer therapies, immunotherapies, cellular, or radiotherapy. No major surgery within 3 weeks prior to first dose of study treatment.
16. Uncontrolled autoimmune hemolytic anemia (AIHA) or immune thrombocytopenia.
17. Consumption of grapefruit, grapefruit products, Seville oranges, or star fruit within 7 days of starting study treatment.
18. Concomitant steroids for disease related pain control are allowed at any dose but must be discontinued prior to any study treatment initiation. Chronic use of corticosteroids is allowed up to ≤ 20 mg prednisone daily for non-cancer related conditions at the time of study start.
19. History of allogeneic or autologous stem cell transplant (SCT) or CAR-T therapy within the last 30 days or with any of the following:
20. Active graft versus host disease (GVHD)
21. Cytopenias from incomplete blood cell count recovery post-transplant;
22. Need for anti-cytokine therapy for residual symptoms of neurotoxicity > grade 1 from CAR-T therapy;
23. Ongoing immunosuppressive therapy.
24. Known history of human immunodeficiency virus (HIV) serum positivity.
25. Active hepatitis B/C.
26. Known central nervous system (CNS) involvement by lymphoma. Patients with previous treatment for CNS involvement who are neurologically stable and without evidence of disease may be eligible if a compelling clinical rationale is provided to sponsor.
27. Known neurologic disorder or residual neurologic toxicities that may put patients at increased risk of neurologic toxicity in the opinion of the investigator.
28. Cardiac abnormalities.
29. Concomitant malignancies or previous malignancies with less than a 1 year disease- free interval at the time of signing consent.
30. A female patient who is pregnant or breast-feeding.
31. Active uncontrolled systemic infection.
32. Received an investigational agent within 30 days or within 5 T1/2, whichever is shorter prior to the first dose of study treatment.
33. Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal (GI) absorption of ibrutinib or venetoclax.
34. Current treatment with certain strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers and/or strong P-gp inhibitors..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Gullbo, MD, Study Director — Theradex Oncology
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No patients were enrolled in Safety Lead-In Cohort 1, Safety Lead-In Cohort 3, and Expansion Phase.
Groups:
- Safety Lead-In Cohort 2: APR-246 + Venetoclax + Rituximab in Subjects with R/R CLL.
  APR-246 (eprenetapopt) + Venetoclax + Rituximab in CLL: APR-246 D1, 8 and 15 of each cycle Venetoclax + Rituximab will be given at a standard dose and schedule
Period: Overall Study
Arm/Group | Safety Lead-In Cohort 2
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Safety Lead-In Cohort 2
Number analyzed (Participants) | 1
Age, Continuous [Median (Full Range); unit: years] | 74 [74 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: To Determine the DLT of APR-246 in Combination With Acalabrutinib or in Combination With Venetoclax + Rituximab Therapy in Subjects With NHL, Including Subjects With R/R CLL, RT and R/R MCL.
Description: The occurrence of DLTs, classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events .
Time Frame: Through study completion, approximately 1 year
Population: Data was not collected as study was terminated.
Arm/Group | Safety Lead-In Cohort 2
Number analyzed (Participants) | 0

2. Primary Outcome: To Assess the Frequency of Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) Related to APR-246 in Combination With Acalabrutinib and With Venetoclax + Rituximab Therapy.
Description: The frequency of TEAEs and SAEs related to APR-246 in combination with acalabrutinib and with venetoclax + rituximab therapy
Time Frame: Through study completion, approximately 6 months
Population: Study was terminated.
Measure: Number; unit: participants
Arm/Group | Safety Lead-In Cohort 2
Number analyzed (Participants) | 1
participants | 1

3. Primary Outcome: To Determine the Maximum Tolerated Dose (MTD) and the Recommended Phase 2 Dose (RP2D) in Subjects With TP53 Mutant NHL, Including Subjects With R/R CLL, RT and R/R MCL.
Description: The highest dose of APR-246 with acceptable toxicity (RP2D of APR-246) (the dose producing ≤ 20% of DLT).
Time Frame: Through study completion, approximately 1 year
Population: Data was not collected as study was terminated.
Arm/Group | Safety Lead-In Cohort 2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: approximately up to 6 months
Description: Study terminated after 1 patient was enrolled in cohort 2. No patients were enrolled in Cohort 1, Cohort 3 and the expansion Phase.
Groups:
- Safety Lead-In Cohort 1: APR-246 + Acalabrutinib in Subjects with R/R CLL.
  APR-246 (eprenetapopt) + Acalabrutinib in CLL: APR-246 D1, 8 and 15 of each cycle Acalabrutinib will be given at a standard dose and schedule
- Expansion Cohorts: APR-246 + (Acalabrutinib, OR, (Ven+R)) in Subjects with R/R TP53-mutant CLL, and/or MCL, and/or RT
  APR-246 (eprenetapopt) + (Acalabrutinib, OR, (Venetoclax +Rituximab)), in CLL and/or MCL and/or RT: APR-246 D1, 8 and 15 of each cycle Acalabrutinib will be given at a standard dose and schedule Venetoclax and Rituxiab will be given at a standard dose and schedule
- Safety Lead-In Cohort 3: APR-246 + Venetoclax + Rituximab in Subjects with RT
  APR-246 (eprenetapopt) + Venetoclax + Rituximab in RT: APR-246 D1, 8 and 15 of each cycle Venetoclax + Rituximab will be given at a standard dose and schedule
Arm/Group | Safety Lead-In Cohort 1 | Safety Lead-In Cohort 2 | Expansion Cohorts | Safety Lead-In Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1 | 0/0 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Lead-In Cohort 1 (N=0) | Safety Lead-In Cohort 2 (N=1) | Expansion Cohorts (N=0) | Safety Lead-In Cohort 3 (N=0)
Dizziness (Nervous system disorders) | NA | 1 (3) | NA | NA
Blood Bilirubin Increased (Investigations) | NA | 1 (4) | NA | NA
Bursitis (Musculoskeletal and connective tissue disorders) | NA | 1 | NA | NA
Constipation (Gastrointestinal disorders) | NA | 1 | NA | NA
Odema Peripheral (General disorders) | NA | 1 | NA | NA
Hyperphosphatemia (General disorders) | NA | 1 | NA | NA
Insomnia (Psychiatric disorders) | NA | 1 | NA | NA
Muscular Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | NA | 1 | NA | NA
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | NA | 1 | NA | NA
Pain (General disorders) | NA | 1 | NA | NA
Vomiting (Gastrointestinal disorders) | NA | 1 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/89/NCT04419389/Prot_SAP_000.pdf